CLINICAL TRIAL: NCT04737265
Title: A Randomized, Open Label Pilot Trial of a Biomarker Guided Strategy of Cardioprotection in Patients With Lymphoma or Breast Cancer Treated With Anthracyclines
Brief Title: Pilot Study of an NTproBNP Guided Strategy of Cardioprotection
Acronym: NTproBNP-Guide
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UPCC 25920; R21HL152148 (NIH)
Record Dates: First submitted 2021-01-28; First posted 2021-02-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Cardiotoxicity; Toxicity Due to Chemotherapy; Breast Cancer; Lymphoma; Cardiomyopathies; Heart Failure
Keywords: Risk-Guided Intervention; Cardiotoxicity of Chemotherapy; Cardio-Oncology; Cardiomyopathy
MeSH Terms: conditions — Cardiotoxicity; Breast Neoplasms; Lymphoma; Cardiomyopathies; Heart Failure

STUDY DESIGN:
Intervention Model Description: Serial monitoring of NTproBNP during chemotherapy will be used to identify high-risk patients in the intervention arm; patients who experience elevations in NTproBNP will be initiated and titrated on a personalized regimen of neurohormonal antagonists. Patients in the usual care arm will not have serial NTproBNP monitoring and will be managed according to usual care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Biomarker Guided Arm (Experimental): NTproBNP will be monitored serially prior to start of anthracycline based chemotherapy, at each cycle of anthracycline based chemotherapy, and at 3 month intervals for a total of 12 months.
  Clinical, echocardiographic, and biomarker data will be collected on all patients at baseline and at standardized intervals at 3, 6, 9, and 12 months following initiation of Anthracycline chemotherapy.
  Interventions: Other: Biomarker Guided Intervention
- Usual Care (No Intervention): NTproBNP will not be monitored while patients are on study unless clinically indicated. Clinical, echocardiographic, and biomarker data will be collected on all patients at baseline and at standardized intervals at 3, 6, 9, and 12 months following initiation of Anthracycline chemotherapy. Biomarker data will also be collected at each cycle of Anthracycline chemotherapy.

INTERVENTIONS:
Other: Biomarker Guided Intervention — NTproBNP above the upper limit of normal will trigger the initiation of heart failure therapy with counseling from a study investigator based on protocol specified algorithm.
  Arms: Biomarker Guided Arm

SUMMARY:
Investigators will evaluate the safety and feasibility of a biomarker-guided cardioprotection strategy using NTproBNP, as compared to usual care, in breast cancer and lymphoma patients treated with anthracyclines.

DETAILED DESCRIPTION:
This is a randomized, open-label pilot trial of a biomarker-guided strategy using NT-proBNP to identify and treat patients with a high risk of cancer therapy-related cardiotoxicity. Patients will be enrolled and randomized prior to initiation of anthracycline-based therapy and followed for 12 months with blood samples, echocardiography, and patient reported outcomes surveys. The overall hypothesis is that a biomarker guided treatment strategy that initiates neurohormonal antagonists in breast cancer or lymphoma patients who have increases in NT-proBNP prior to, during, or after anthracyclines will be feasible, well-tolerated, and result in attenuation of cardiotoxicity, compared to standard care.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent and HIPAA authorization
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, ≥ 18 years of age
* Diagnosed with breast cancer or lymphoma (any subtype), planned to receive an anthracycline based chemotherapy regimen. Patients may be enrolled up to their first dose of anthracycline even if they have already received other chemotherapeutic or targeted agents as part of neo-adjuvant or adjuvant systemic therapy.

Exclusion Criteria:

* Diagnosed with Stage IV breast cancer
* Uncontrolled blood pressure defined by SBP > 180mmHg on two or more occasions and taking three or more antihypertensives within 1 month prior to enrollment.
* Baseline systolic blood pressure < 90mmHg within 1 month prior to enrollment (if multiple blood pressures are available in the medical record within 1 month prior to enrollment, the average SBP will be considered)
* Women must not be pregnant or breast-feeding due to the potential harm to an unborn fetus and possible risk for adverse events in nursing infants with some anti-hypertensives, including angiotensin receptor blockers. All females of childbearing potential must have a blood test or urine study within 10 days prior to enrollment to rule out pregnancy. All females of childbearing potential must be strongly advised to use accepted and effective methods of contraception or to abstain from sexual intercourse for the duration of their participation in the study. A female of childbearing potential is defined as any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
* Patient with prior or concurrent malignancy whose natural history of treatment, in the opinion of the investigator, has the potential to interfere with the safety or efficacy assessment of the investigational regimen
* Patient must not have any of the following
* Severe hepatic impairment, defined as serum bilirubin > ULN, or AST or ALT > 5.0 ULN on most recent labs prior to enrollment. Results of serum bilirubin, AST, and ALT must be checked for screening if no results available in the EMR within 28 days prior to enrollment.
* end-stage renal failure on dialysis
* hyperkalemia with a potassium > 5.5 mEq/l on most recent labs prior to enrollment. Serum potassium must be checked for screening if no results available in the EMR within 28 days prior to enrollment.
* a history of kidney transplant
* an eGFR < 30 ml/min/1.73m2 at most recent check prior to enrollment. Creatinine must be checked for screening if no results available in the EMR within 28 days prior to enrollment
* cardiogenic shock
* decompensated heart failure requiring the use of IV inotropic therapy
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
Recruitment Rate | At baseline
  percent of eligible patients who are randomized
Retention rate | Through study completion (expected to be 1 year)
  percent of randomized patients who complete the study per protocol
Adherence rate | Through study completion (expected to be 1 year)
  percent of study activities completed in window
Compliance rate | Through study completion (expected to be 1 year)
  Compliance by PROMIS Scale v1.0 for patients in the biomarker guided arm initiated on heart failure medications
Maximum tolerated dose | Through study completion (expected to be 1 year)
  Maximum tolerated dosage of neurohormonal antagonist medications for patients in the biomarker-guided arm with NTproBNP above upper limit of normal
Incidence of Adverse Events | 12 months
  Rate of Grade 2 or higher adverse events by CTCAEv5.0

SECONDARY OUTCOMES:
Change in NTproBNP | Through study completion (expected to be 1 year)
  Change in clinically measured NTproBNP following initiation of neurohormonal antagonists in patients with NTproBNP above upper limit of normal in the biomarker guided arm
Change in Left ventricular ejection fraction (LVEF) by Echocardiogram | 12 months
  Change in core-lab quantitated left ventricular ejection fraction
Incidence of cardiotoxicity | 12 months
  Incidence of cardiotoxicity defined as LVEF decline of at least 10% to less than 50%
Incidence of Hear Failure (HF) | 12 months
  Incidence of new or worsened clinical heart failure, defined as urgent or new office or emergency department visit or hospitalization for HF, adjudicated by a clinical events committee
Frequency of cancer treatment interruptions | Through study completion (expected to be 1 year)
  Frequency of cancer treatment interruptions due to cardiotoxicity

OTHER OUTCOMES:
Change in diastolic function on echo | 12 months
  Change in E/e' by echo
Change in longitudinal strain | 12 months
  Change in global longitudinal strain by echocardiogram
Change in circumferential strain | 12 months
  Change in circumferential strain by echocardiogram
Change in high sensitivity troponin (hsTnT) | 12 months
  Change in hsTnT measured in batches from banked samples
Change in Growth Differentiation Factor 15 (GDF-15) | 12 months
  Change in GDF-15 measured in batches from banked samples
Change in myeloperoxidase (MPO) | 12 months
  Change in MPO measured in batches from banked samples
Change in NTproBNP (post hoc batch analysis) | 12 months
  Change in NTproBNP measured in batches from banked samples for all patients on both arms
Change in patient reported activity level | 12 months
  Change in total weekly leisure activity in METS (assessed by GODIN Leisure Time Exercise Questionnaire)
Change in patient reported symptoms | 12 months
  Change in MD Anderson Symptoms Inventory - Heart Failure (MDASI-HF). Higher scores indicate increased symptom severity or symptom distress.
Change in patient reported fatigue | 12 months
  Change in Patient Reported Outomes Information System (PROMIS) Fatigue Score. A higher score corresponds to higher levels of reported fatigue.
Change in patient reported quality of life | 12 months
  Change in Patient Reported Outomes Information System (PROMIS) Global Health score. Higher scores indicate a healthier patient.
Change in patient reported adverse events | 12 months
  Change in NCI Patient Reported Outcomes - Common Terms and Criteria for Adverse Events (PRO CTCAE).
Incidence of treatment interruptions in administration of anthracycline chemotherapy | 12 months
  Incidence of anthracycline chemotherapy being held or discontinued secondary to side effects or toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Ky, MD, MSCE, Principal Investigator — Perelman School of Medicine at the University of Pennsylvania
Locations (3):
- United States (3):
  - City of Hope, Duarte, California
  - Abramson Cancer Center at University of Pennsylvania, Philadelphia, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Xia C, Smith AM, Lefebvre B, Jamal FA, Armenian SH, Koropeckyj-Cox D, Zhang L, Liu PP, Landsburg D, Clark AS, Shah PD, Hubbard RA, Huang A, Golec S, Hewitt M, Wilcox NS, Chen Z, Rethy L, Jung W, Ko K, Narayan V, Martei YM, Lang NN, Januzzi JL, Felker GM, Ky B. Biomarker-Guided Cardioprotection for Patients Treated With Anthracyclines: A Randomized Clinical Trial. JAMA Netw Open. 2025 Dec 1;8(12):e2546201. doi: 10.1001/jamanetworkopen.2025.46201. PMID 41335439